CLINICAL TRIAL: NCT06116747
Title: Strengthening First-time Fathers' Engagement in Early Parenthood When Having a Preterm Infant - The SUPPORTED Study.
Brief Title: The SUPPORTED Study - First-time Fathers of Preterm Infants.
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Collaborators: Odense University Hospital (Other); Rigshospitalet, Denmark (Other); Holbaek Sygehus (Other); Slagelse Hospital (Other); Zealand University Hospital (Other); Gødstrup Hospital (Other); Aarhus University Hospital (Other); Aalborg University Hospital (Other); University College Absalon (Other); Lovisenberg Diakonale Hospital (Other)
Responsible Party: Principal Investigator, Anne Brodsgaard, Professor, Hvidovre University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: P-2022-792
Record Dates: First submitted 2023-10-31; First posted 2023-11-03 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Preterm; Father-Child Relations
Keywords: Preterm; Father-Child relations
MeSH Terms: conditions — Premature Birth | interventions — Methods

STUDY DESIGN:
Intervention Model Description: Intervention study with one control group and one intervention group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No intervention Group (No Intervention): Group receiving care as usual
- Intervention Group (Experimental): Complex Intervention under development in collaboration with fathers' health care professionals in primary and secondary sectors.
  Interventions: Behavioral: Intervention

INTERVENTIONS:
Behavioral: Intervention — Support for fathers of preterm infants
  Arms: Intervention Group

SUMMARY:
The purpose is to support first-time fathers of premature infants in early parenthood by promoting early paternal-infant relationships. Improve paternal confidence by involving, knowledge sharing, and guiding them in their premature infants' emotional, nutritional, and developmental needs.

The study operates with two study populations: a) first-time fathers, their premature infants, and families, b) health care professionals working with new families in neonatal intensive care units and maternity units and the families' health visitors from the secondary health care sectors. Seven hospitals located in Denmark's five regions participates.

Four studies address the key questions for the father's involvement in supportive health care: 1) How do fathers experience their participation in father-groups in the NICU, 2) What are the first-time fathers' needs and preferences for supporting health care, 3) Development of an intervention based on the identified need to support the fathers in early parenting, 4) Study the process and effect of the intervention on paternal confidence and stress.

The first question is explored in a qualitative evaluation of an ongoing father-group intervention in a neonatal intensive care unit. The following three questions are studied through an action research approach, identifying first-time fathers' needs for support and the current practices among health professionals towards new first-time fathers of premature infants. Secondly, developing guiding principles for health care professionals to strengthen fathers' partnership in health care. Finally, conducting a quasi-experimental study to evaluate the process and effect of the proposed approaches. The study of this paternal supportive programme, involves perspectives that have not yet been studied in Denmark or internationally.

DETAILED DESCRIPTION:
Project description The overall aim of this research study is to identify, develop and evaluate whether supportive strategies for first-time fathers (FTF) of preterm infants will improve parental confidence, mood and anxiety as well as increasing paternal reflective function, and improve infants social-emotional competencies during admission in the Neonatal Intensive Care Unit (NICU), or Maternity Unit (MU) and follow up at home by health visitors in the municipalities in all five regions in Denmark. Thus, improve paternal confidence in the father role by involving, knowledge sharing, and guiding them in their infants' emotional, nutritional, and developmental needs.

Background Developing paternal confidence and engaging in the paternal role is pivotal to men's transition into fatherhood (1). The change in fatherhood culture from breadwinner to being involved in the care of the infant is challenging (2-4). Among first-time parents, fathers express more insecurity than mothers (5). Fathers of preterm infants experience even more insecurity as it is more difficult to read the infant's cues (6). Fathers have unique support needs that are frequently unmet (5,7), which may result in decreased mental health, father-infant interaction, and parenting confidence (7). In the health care system, they often feel like bystanders (4) even though they want a participating role to attach to the infant (8).

In Denmark, about 4.200 of 60.000 infants (7%) are born preterm (9). Preterm infants are admitted to the hospital for weeks or months due to immaturity of the organs. Information, emotional and practical support from healthcare professionals (HCP) are needed to enhance parents' experiences, well-being, caring, and confidence during admission and at home (10). Studies on fathers' involvement in early interventions of their preterm infant are limited (11). Generally, interventions that extend over a long period of time and include both primary and secondary sectors are the most effective (12). Studies have addressed parental relationships and insecurity and sought interventions to improve parents' opportunities to actively participate in care, showing positive effects, e.g., skin-to-skin helps fathers gain confidence in the paternal role (13). Across sections nurses, midwives, and health visitors provide early parenting support to all new families. There is a need to change the culture among HCP to increase the engagement of the father in a family-focused approach, and this requires the identification of changeable factors among HCPs in primary and secondary sectors like knowledge, attitudes, and behavior (14). Perceptions of fathers as important as the mother in early parenting are associated with favorable attitudes toward including them in family interventions; this association is mediated by the professionals' perception of their confidence (15).

Health- and socio-economic arguments exist for improving early paternal engagement, and fathers want to be engaged, attentive, and caring (16). Their involvement in fatherhood can benefit the health and well-being of both himself, the mother, and the infant (17). Fathers' engagement has been shown to improve social and relational functioning in childhood, decrease behavioral problems in adolescence, and increase educational outcomes (18,19).

Even though the Nordic countries have been at the forefront of involving fathers in pregnancy and delivery, evidence shows that fathers are still not included and approached by HCP equally to mothers. This project which works at and within all levels in the healthcare sector and across the country, has the potential to take the next step to a partnership with FTF of preterm infants by changing practice and culture to benefit the fathers, preterm infants, and families.

Setting, recruitment and participants The recruitment period of first-time fathers and their partners starts November 6th 2023 and is expected to be completed late July 2027 by health professionals at the NICU in participating hospital settings in all Danish regions where preterm infants are admitted. Eligible yearly from hospitals of Aalborg/Gødstrup (n=150), Aarhus (n=155), Odense (n=80), Slagelse (n=75), Holbæk (n=50), Roskilde (n= 80), Rigshospitalet (n=140) and Hvidover (n=170), and municipalities in the hospitals' catchment areas. About 40% are FTFs, and about 12% not fulfilling the inclusion criteria. When a total of 900 families will be eligible yearly there is a good possibility to recruit 266 families in both groups in the recruitment period. Eight hospitals representing all Regions in Denmark and municipalities in their catchment areas will participate.

The primary study population consists of FTF and their preterm infants (i.e., infants born alive before 37 weeks of pregnancy). Inclusion criteria: Danish-speaking FTF to preterm infants admitted to a NICU. Exclusion criteria: parents unable to manage their own legal affairs and not living at home. The secondary study population consists of nurses and midwives at hospitals and health visitors in the municipalities. For the time and activity schedule (see appendix 1).

Framework This project will use the Medical Research Councils' (MRC) framework for developing and evaluating complex interventions as the overall frame of reference (20), including developing, feasibility testing, implementing, and evaluating the intervention. This national study comprises three interlinked studies, including an intended and beneficial collaboration between FTF and HCP across sectors from the NICU and health visitors from the municipalities. The project may promote a joint responsibility agreement between health care providers from municipalities and hospitals with the aim to promote knowledge and skills across sectors about caring for new family with preterm infants. New knowledge and skills might promote both groups confidence and motivation working with first-time fathers of preterm infants. Each study forms the foundation of the following study that ensures a constant focus on the context, existing practice, and feasibility of the planned study activities.

STUDY 1 - THE ASSESSMENT PHASE AND STUDY 2 - THE DEVELOPMENTAL PHASE We expect the intervention to be supported by technology and to include a training program for HCPs describing how to deliver the intervention as intended. The training program is expected to include a) an implementation manual, b) e-learning and face-to-face training, and c) supervision workshops. Based on prior studies (13,31,32), the intervention for fathers is expected to contain; a) Guidance in understanding the infant's strengths and needs concerning care, feeding, sleeping, and comfort; b) support to build a healthy father-infant relationship and c) strengthening of fathers in being fathers while supporting the mothers. However, this will be elucidated and adjusted according to pilot testing and the findings of studies 1 and 2.

STUDY 3 - THE IMPLEMENTATION AND EVALUATION PHASE Implementation and evaluation of the developed intervention. The content and format of the intervention is shaped by the outcomes of study 1 and 2.

Aim The aim is to explore whether the intervention has positive effects on fathers and infants' well-being and to unfold barriers and facilitators of the implementation through process evaluation.

Implementation and evaluation The manual for the HCP from municipalities and hospitals, the training course, and the supervision workshop during the intervention period ensure that both sectors deliver the program as intended.

The effect evaluation explores whether the intervention has positive effects on the father and the infant and thereby determines the success of the project. We hypothesize that a tailored intervention, developed according to the identified needs, will increase paternal confidence and mood and reduce anxiety and stress. Moreover, it will increase the father's capacity to mentalize in the early father-infant relationship, improve the infant's socio-emotional behavior, as well as increase exclusive breastfeeding rates at two weeks and four months of corrected age. Parallel to the effect evaluation a process evaluation will be conducted with the aim to evaluate fathers' and health professionals' experiences with the study. Furthermore, to determine whether the project has been implemented as intended.

Methods An effect evaluation of the intervention will be performed in a quasi-experimental design with the following outcome measures: Primary outcome: Paternal confidence (KPCS) (33,34). Secondary outcomes: Family assessment (FAD) (35,36). Paternal stress scale (37,38), reflective functioning (PRFQ) (39), depressive symptoms (GS) (40), and child social and emotional development (ASQ:SE) (41). We also collect data from the mothers to make sure that increased focus on the father does not negatively impact her. Data on the comparison group will be collected alongside the development of the intervention to avoid spillover effects.

Sample size The power calculation is based on the primary outcome. Instruments measuring early confidence concerning early fatherhood are unknown. Twenty-five percent of new mothers have a risk score <37 on the KPCS scale. First-time fathers have been shown to be more insecure than new mothers (39,40). We estimate that 60% of first-time fathers to preterm infants have a risk score <37 on the KPCS scale. With a significance level of 5% and a power of 80%, the power calculation finds a need for 173 participating first-time fathers in each group to be able to identify a statistically significant difference decrease of 15% in reporting low confidence as a father. To be able to account for potential confounders (age, marital status, educational background, and employment), 10 fathers will be added per confounder giving 213 in each group. Additionally, accounting for the expected loss to follow up of 20 % gives a final need of 266 fathers in each group.

Statistical methods The effect of the intervention on the primary outcome, paternal confidence scale, will be analyzed by chi-squared test on distribution for <37 and ≥37 between intervention and comparison groups. To evaluate possible confounders, a logistic regression model will be used. If the confounding effect is more than 10%, the variable is included in the final model. The secondary outcomes will be compared using a t-test or Wilcoxon rank sum test if normality assumption is not satisfied. Confounders will be evaluated with the same procedure as for KPCS, with linear regression used instead of logistic regression.

Analysis of qualitative data Interview data will be analyzed using systematic text condensation, which consists of four steps: (I) read transcripts repeatedly to identify themes; (II) identify and code units of meaning; (III) identify sub-groups of codes from step II and develop condensates from them; and (IV) describe experiences based on the condensates.

Process evaluation Alongside the effect evaluation, a process evaluation will be conducted to assess the reach, dose, and fidelity of the intervention to unfold facilitators and barriers to implementation as well as the influence of contextual factors.

Ethics Approval from the Danish Committees on Health Research Ethics was not required for this project (journal no.: F-22055527). Permission has been obtained from the Danish Data Protection Agency via Pactius, the Capital Region of Copenhagen (journal no.: P-2022-792). Data will be collected through a REDCap database, and all data will be stored in the hospital server's logged drive. Permission to use the different internationally validated questionnaire scales will be obtained from the copyright holders. According to the Declaration of Helsinki, data will be handled anonymously, and written informed content will be obtained from all participants.

ELIGIBILITY:
Inclusion Criteria:

* First-time fathers of preterm infants
* Co-habitating with the mother of the infant
* Neonatal Admission for more than seven days
* Danish language
* Infants born before the 37 week of gestation

Exclusion Criteria:

* Infant receiving palliative treatment and care
* parents not discharged for home
* parental mental illness

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — First-time fathers and mothers of preterm infants
Enrollment: 532 (Estimated)
Dates: Start 2023-10-31 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Paternal confidence: Karitane Parenting Confidence Scale (KPCS), | 2 weeks, 4 month, 9 month corrected age
  15 items, 0-1 year postpartum. (Črnčec et al., 2008, 2010).

SECONDARY OUTCOMES:
Infant social-emotional competence | 4 month, 9 month corrected age
  Ages and stages questionnaire: Social-Emotional (ASQ:SE). 23 items, 3-9 months postpartum. (Squires et al., 1997).
Depression | 2 weeks, 9 month corrected age
  Gotland Male Depression Scale (GMDS) 13 items. (Sigurdsson et al, 2014).
FAD: Family Assessment Device | 4 month corrected age
  12 items) (Thastum et al 2009, Boterhoven De Haan et al 2015).
Paternal mentalizing competence: The Parental Reflective Functioning Questionnaire (PRFQ) | 4 month corrected age
  18 items, 0-5 years postpartum. (Allen et al., 2008; Slade, 2005; Slade et al., 2005; UCL, 2022). 18 items, 0-5 years postpartum. (Allen et al., 2008; Slade, 2005; Slade et al., 2005; UCL, 2022).
Exclusive breastfeeding direct from the breast (2 items) | 2 weeks, 4 month, 9 moths correced age
  Does the mother of your infant exclusively breastfeed? Yes/no.- If not, when did the mother stop exclusively breastfeeding? (WHO, 2015, 2018, 2022a, 2022b)
Paternaty leave | 4 month and 9 moths corrected age
  (2 items)
PSS: Parental Stress Scale | 2 weeks, 4 month corrected age
  18 items - The items statements are reated for agreement by prants using a 5-point response scale (1=strongly disagree, 2= disagre, 3= undecided, 4= agree, 5= Stongly agree.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Brødsgaard, Principal Investigator — Hvidovre University Hospital
Locations (1):
- Copenhagen University Hospital Amager Hvidovre, Hvidovre, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Holm KG, Hagi-Pedersen MB, Haslund-Thomsen H, Nilsson I, Aagaard H, Maastrup R, Ejlertsen C, Petersen M, Feenstra MM, Kristensen I, Brodsgaard A. Protocol for the SUPPORTED study: a Danish multicentre complex intervention for first-time fathers of preterm infants. BMJ Open. 2025 Sep 15;15(9):e100258. doi: 10.1136/bmjopen-2025-100258. PMID 40954083